CLINICAL TRIAL: NCT05733663
Title: Persistent Increase in the Intestinal γδ+ T-cell Subset: A Potential Biomarker of Coeliac Disease in Patients Started on a Gluten-free Diet
Brief Title: TCRγδ+ Cells After Gluten-free Diet: A Biomarker for Coeliac Disease?
Acronym: GFDL
Status: Completed | Type: Observational
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: GFDL
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Celiac Disease
Keywords: Coeliac disease; Gluten-free diet; Intraepithelial lymphocytes; Villous atrophy
MeSH Terms: conditions — Celiac Disease | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients diagnosed with coeliac disease: A group of paediatric or adult patients diagnosed with CD and started on a strict GFD, with baseline and a follow-up intestinal biopsy to assess histological and intraepithelial lymphogram at least 1-year after starting the GFD, and with increased γδ+ T-cells at baseline.
  Interventions: Diagnostic Test: Endoscopic procedure with duodenal biopsy

INTERVENTIONS:
Diagnostic Test: Endoscopic procedure with duodenal biopsy — * In all patients the investigators will analyse coeliac serology, DQ-genotype, and results of two duodenal biopsy sampling (one at diagnosis before starting the GFD and another sampling during follow-up with GFD) for assessment of both histopathology and intraepithelial lymphocyte subpopulations by T-cell flow cytometry. In addition, clinical, serological, and histological response to GFD will be evaluated.
  * T-cell flow cytometry assay is performed as previously described by our group in previous studies. In all patients, an additional duodenal biopsy sample is taken from the second-third portion of the duodenum at the same endoscopic procedure that for histopathology. The normal cut-off values for the IEL cytometric pattern in our laboratory are CD3+TCRγδ+ IEL ≤8.5% (≤mean + 2SD) and CD3- IEL ≥10% (10th percentile). The cut-offs define four intraepithelial lymphogram patterns: normal, isolated decrease in CD3- cells, isolated increase in TCRγδ+ cells, and the coeliac lymphogram.

SUMMARY:
Coeliac disease (CD) is a systemic process of autoimmune nature related to the existence of a permanent intolerance to gluten and manifests itself in genetically susceptible individuals. It has a global prevalence of 0.5-1.5%. The diagnosis of CD should be made in patients following a normal gluten-containing diet and is based on coeliac serology and histopathological changes of the small intestinal mucosa. However, nowadays many patients come to their doctor to rule out CD after having started a gluten-free diet (GFD) with improvement of symptoms. In this scenario, making the diagnosis of CD remains a challenge, as it must be considered that most CD-associated changes revert after gluten withdrawal.

An essential finding of CD is the increased number in total intraepithelial lymphocytes (IEL) in the duodenal mucosa, later characterized by an expansion of γδ+ and CD8+ IEL coupled to a decrease in CD3- IEL. An accurate quantification of the γδ+ subset became possible with the introduction of flow cytometry. In 2002, Spanish investigators proposed a diagnostic algorithm for paediatric CD that included the combined use of a high percentage of γδ+ and a low percentage of CD3- IEL, which was termed the coeliac lymphogram, which has been shown to be very accurate for the diagnosis of CD. Thus, the use of flow cytometric phenotyping of IEL may strengthen the diagnosis of CD when it is not straightforward.

This study will provide information about the potential usefulness of T-cell flow cytometric coeliac patterns as CD biomarkers to confirm the diagnosis of CD in patients who have already started a GFD. These results may help to make decisions in specific situations of routine clinical practice, avoiding bothersome gluten reintroduction and delays in diagnosis.

DETAILED DESCRIPTION:
Hypothesis:

The increase in the TCRγδ+ subset appears to be permanent despite a GFD, which opens up the possibility of using it as a diagnostic tool in patients following a GFD, without the need to undergo gluten challenge. Several studies have focused on this aspect with promising results, but the studies have been performed on small samples of patients, and follow-up time after a GFD has not always been described or only changes in mean values before versus after the diet have been reported.

ELIGIBILITY:
Inclusion criteria:

* Paediatric or adult patients diagnosed with CD and started on a strict GFD
* Patients with a follow-up intestinal biopsy to assess histological remission at least 1-year after starting the GFD
* Assessment of the intraepithelial lymphogram at both baseline and follow-up
* Presence of increased TCRγδ+ cells at baseline.

Exclusion criteria:

* Refusal of the patient to participate in the registry.
* Pregnancy and severe comorbidities (heart disease, chronic obstructive pulmonary disease, liver disease, bleeding disorders, etc).
* Patients with intake of NSAIDs or Olmesartan.
* Patients with Crohn's disease, autoimmune disease associated enteropathy, collagenous sprue, microscopic colitis, lymphocytic enteritis due to intestinal parasitosis or Helicobacter pylori infection, other enteropathies.
* Selective IgA deficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * All patients included in the 'Prospective hospital registry of patients with suspected coeliac disease', who fulfil the inclusion criteria and none of the exclusion criteria in present study.
  * Study period: The study period will be 8 years (January 2013 - December 2020).
  * Diagnosis of CD will be based on the 2019-guidelines of the European Society for the Study of Coeliac Disease, and the recent Paris consensus criteria about diagnosis of seronegative CD. Presence of a compatible T-cell flow cytometric coeliac pattern will be considered as complementary for diagnosis of seronegative CD.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of long-term persistence of both the coeliac lymphogram (increase in TCRγδ+ and decrease in CD3- cells) and the isolated increase in TCRγδ+ cells measured by T-cell flow cytometry in CD patients after starting a GFD. | 1 year
  Lymphocyte subpopulations (TCRγδ+ and CD3- cells) are measured by flow cytometry.

SECONDARY OUTCOMES:
Percentage of loss of the T-cell flow cytometric coeliac pattern (increase in TCRγδ+) according to baseline histology (measured by Marsh Classification: 0, 1, 2 or 3) | 1 year
  To assess the frequency of nonpersistence of the increased TCRγδ+ subset related to study variables, the chi-square test, Fisher exact test, and the Freeman-Halton extension of the Fisher exact probability test for a 2x3 or a 2x4 contingency table were used.
Percentage of loss of the T-cell flow cytometric coeliac pattern (increase in TCRγδ+) according to age group (measured by years). | 1 year
  To assess the frequency of nonpersistence of the increased TCRγδ+ subset related to study variables, the chi-square test, Fisher exact test, and the Freeman-Halton extension of the Fisher exact probability test for a 2x3 or a 2x4 contingency table were used.
Percentage of loss of the T-cell flow cytometric coeliac pattern (increase in TCRγδ+) according to gender (classified according to male or female sex). | 1 year
  To assess the frequency of nonpersistence of the increased TCRγδ+ subset related to study variables, the chi-square test, Fisher exact test, and the Freeman-Halton extension of the Fisher exact probability test for a 2x3 or a 2x4 contingency table were used.
Percentage of loss of the T-cell flow cytometric coeliac pattern (increase in TCRγδ+) according to coeliac serology (measured by presence or absence of anti-transglutaminase antibodies). | 1 year
  To assess the frequency of nonpersistence of the increased TCRγδ+ subset related to study variables, the chi-square test, Fisher exact test, and the Freeman-Halton extension of the Fisher exact probability test for a 2x3 or a 2x4 contingency table were used.
Percentage of loss of the T-cell flow cytometric coeliac pattern (increase in TCRγδ+) according to DQ-genotype (measured by presence or absence of HLA-DQ2.5). | 1 year
  To assess the frequency of nonpersistence of the increased TCRγδ+ subset related to study variables, the chi-square test, Fisher exact test, and the Freeman-Halton extension of the Fisher exact probability test for a 2x3 or a 2x4 contingency table were used.
Percentage of loss of the T-cell flow cytometric coeliac pattern (increase in TCRγδ+) according to follow-up time (measured by years). | 1 year
  To assess the frequency of nonpersistence of the increased TCRγδ+ subset related to study variables, the chi-square test, Fisher exact test, and the Freeman-Halton extension of the Fisher exact probability test for a 2x3 or a 2x4 contingency table were used.

OTHER OUTCOMES:
Frequency of persisting CD changes despite a GFD (i.e., positive CD serology, persistent villous atrophy) at the time of follow-up biopsy and compare them with the frequency of a persistent increase in γδ+ subset. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maria Esteve, PhD, MD, Principal Investigator — Hospital Universitari Mútua Terrassa
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No